CLINICAL TRIAL: NCT02635724
Title: A Phase 3, Multicenter, Single-arm, Open-label, Study to Evaluate the Safety, Pharmacokinetics and Effectiveness of Intravenous Peramivir in Elderly Subjects With Acute Uncomplicated Influenza Infection and in Subjects With Acute Uncomplicated Influenza Infection at Higher Risk for Influenza Complications
Brief Title: Safety, PK and Effectiveness of IV Peramivir in Elderly and Higher Risk Subjects With Uncomplicated Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX1812-306
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Influenza
Keywords: Acute uncomplicated; Elderly
MeSH Terms: conditions — Influenza, Human | interventions — peramivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peramivir (Experimental): Single dose 600 mg IV injection
  Interventions: Drug: Peramivir

INTERVENTIONS:
Drug: Peramivir
  Other Names: Rapivab

SUMMARY:
This study will evaluate the safety, pharmacokinetics and effectiveness of a single dose of 600 mg IV peramivir in the treatment of elderly subjects with acute uncomplicated influenza infection and in subjects with acute uncomplicated influenza infection at higher risk for influenza complications. All subjects will receive IV peramivir.

ELIGIBILITY:
Inclusion Criteria:

* A positive influenza Rapid Antigen Test (RAT) and/or a FDA-approved PCR test and at least one clinical sign or symptom consistent with acute influenza infection as listed below OR
* Clinical signs and symptoms consistent with acute influenza infection consisting of an oral temperature ≥ 100°F (37.8°C) with at least one respiratory symptom of at least moderate severity (cough or rhinitis) and at least one constitutional symptom of at least moderate severity (myalgia [aches and pains], headache, feverishness, or fatigue)
* Influenza symptom onset < 48 hours. However, due to historically delayed presentation for medical care in the adult population, approximately 20% of the elderly population may be enrolled with symptoms starting > 48-hours but ≤ 72-hours

Exclusion Criteria:

* Women who plan to breast-feed for the first 48 hours after study drug administration
* Subjects requiring hospital admission to treat medical condition(s) which could represent complications of influenza.
* Recent worsening of any chronic medical condition consistent with complications of influenza
* Current evidence of a bacterial infection requiring antibiotic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-12; Primary Completion 2018-04 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Clark, MD, Principal Investigator — Prof., Dept. of Emergency Medicine, Oakland University, William Beaumont School of Medicine, Royal Oak, MI
Locations (15):
- United States (15):
  - Peramivir Investigational Site, Brooksville, Florida
  - Peramivir Investigational Site, Lakeland, Florida
  - Peramivir Investigational Site, Miami, Florida
  - Peramivir Investigational Site, St. Petersburg, Florida
  - Peramivir Investigational Site, Tampa, Florida
  - Peramivir investigative site, Indianapolis, Indiana
  - Peramivir investigative site, Detroit, Michigan
  - Peramivir Investigational Site, Dayton, Ohio
  - Peramivir investigative site, Smithfield, Pennsylvania
  - Peramivir Investigational Site, Houston, Texas
  - Peramivir Investigative Site, San Antonio, Texas
  - Peramivir investigative site, Splendora, Texas
  - Peramivir Investigational Site, Draper, Utah
  - Peramivir Investigational Site, Salt Lake City, Utah
  - Peramivir investigative site, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A single dose of IV peramivir was administered to elderly subjects (≥ 65 years old) and at risk subjects with acute uncomplicated influenza. Subjects received a single IV dose of 600 mg peramivir if they had creatinine clearance (CLCR) ≥ 50 mL/min and a reduced dose if they had CLCR < 50 mL/min (200 mg for CLCR 30 to 49 mL/min and 100 mg for CLCR 10 to 29 mL/min).
Groups:
- At Risk (<65 Years): A single IV dose of peramivir was administered to adults considered at risk, including pregnant women, residents of long-term care facilities, American Indians and Alaskan Natives, as well as those with comorbidities (e.g. asthma, heart disease, diabetes) that increased the risk of complications.
- Elderly (65-75 Years): A single IV dose of peramivir was administered to adults aged 65 to 75 years
- Very Elderly (>75 Years): A single IV dose of peramivir was administered to adults aged over 75 years
Period: Overall Study
Arm/Group | At Risk (<65 Years) | Elderly (65-75 Years) | Very Elderly (>75 Years)
Started | 41 | 26 | 7
ITT Population (Intent-to-Treat (ITT) population included all enrolled subjects.) | 41 | 26 | 7
Safety Population (The safety population included all enrolled subjects who received any amount of study drug.) | 41 | 25 | 7
ITTI Population (Intent-to-Treat Infected (ITTI) population included all subjects who were enrolled, treated, and had influenza type A or B confirmed by PCR.) | 28 | 19 | 5
E-R Population (Exposure-Response (E-R) population included all subjects in the ITTI population who had a quantifiable peramivir concentration on Day 1 and had at least one post-baseline effectiveness assessment.) | 28 | 19 | 5
Completed | 41 | 25 | 7
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- At Risk (<65 Years): A single IV dose of peramivir was administered to adults considered at risk
- Total: Total of all reporting groups
Arm/Group | At Risk (<65 Years) | Elderly (65-75 Years) | Very Elderly (>75 Years) | Total
Number analyzed (Participants) | 41 | 25 | 7 | 73
Age, Continuous [Mean (Standard Deviation); unit: Age at screening (years)] | 43.1 (10.67) | 68.4 (3.10) | 81.1 (3.03) | 55.4 (16.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 20 | 4 | 53
  Male | 12 | 5 | 3 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 4
  White | 37 | 23 | 7 | 67
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Baseline Influenza Viral Titre [Number; unit: participants]
  Positive | 27 | 15 | 2 | 44
  Negative | 12 | 3 | 3 | 18
  Missing | 2 | 7 | 2 | 11
Baseline Temperature Status [Number; unit: participants]
  Normal | 16 | 9 | 5 | 30
  Fever | 25 | 16 | 2 | 43
Baseline Composite Influenza Symptom Score [Mean (Standard Deviation); unit: Composite Influenza Symptom Score] — Subjects were asked to provide an assessment of 7 influenza symptoms (cough, sore throat, nasal congestion, myalgia [aches and pains], headache, feverishness, and fatigue) on a 4-point severity scale (0, absent; 1, mild; 2, moderate; 3, severe). Baseline Composite Symptom Score is defined as the sum of the symptoms of influenza recorded by the subject in the diary prior to the initiation of study drug. The maximum possible score is 21.
  Composite Influenza Symptom Score | 14 (3.4) | 15 (3.0) | 10 (5.1) | 14 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability, as Measured by the Number of Adverse Events.
Description: Safety was evaluated through assessment of Adverse Events (AEs).
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | At Risk (<65 Years) | Elderly (65-75 Years) | Very Elderly (>75 Years)
Number analyzed (Participants) | 41 | 25 | 7
Participants
  Subjects with at Least 1 Adverse Event | 17 | 9 | 1
  Subjects with at Least 1 Adverse Event Related to Study Drug | 5 | 3 | 0
  Subjects with at Least 1 Adverse Event Leading to Study Discontinuation | 0 | 0 | 0
  Subjects with at Least 1 Severe or Life-Threatening Adverse Event | 0 | 1 | 0
  Subjects with at Least 1 Severe or Life-Threatening Adverse Event Related to Study Drug | 0 | 0 | 0

2. Secondary Outcome: Plasma Exposure of IV Peramivir as Measured by Drug Concentrations up to 3 Hours Post Infusion
Description: Up to 3 plasma samples will be drawn, where possible: immediately following infusion, 30 mins to 1 hr post-infusion & 1 to 3 hrs post-infusion. Maximum concentration (Cmax), area under the concentration vs. time curve (AUC) from time 0 to 1 hour (AUC0-1), AUC from time 0 to 1.5 hours (AUC0-1.5), and AUC from time 0 to the last measurable time point (AUC0-last) were calculated in Phoenix® WinNonlin® v6.4. No summary statistics were reported due to the variation in the infusion time and sampling times.
Time Frame: up to 3 hours post peramivir infusion
Population: 73 subjects from the ITT population had sufficient PK samples collected for inclusion in the peramivir PK analysis
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | At Risk (<65 Years) | Elderly (65-75 Years) | Very Elderly (>75 Years)
Number analyzed (Participants) | 41 | 25 | 7
h*ng/mL
  AUC0-last | 42400 (15630) | 68300 (116800) | 64600 (66380)
  AUC0-1: number analyzed (Participants) | 41 | 24 | 7
  AUC0-1 | 30600 (15260) | 53600 (107400) | 54400 (63620)
  AUC0-1.5: number analyzed (Participants) | 20 | 12 | 1
  AUC0-1.5 | 38200 (12800) | 85800 (168000) | 35000 (0)

3. Secondary Outcome: Time to Resolution of Fever
Description: Time for fever resolution based on subject diary record of temperature recorded twice daily. A subject had resolution of fever if he/she had an oral temperature < 37.4°C/99.4°F oral and no antipyretic medications were taken for at least 12 hours. The time to resolution of fever was estimated for each age group and overall using the Kaplan-Meier method with temperature and symptom relief medication information obtained from the Subject Diary data. Subjects who did not have resolution of fever were censored at the time of their last non-missing post-baseline temperature assessment.
Time Frame: 14 days
Population: Intent to treat infected (ITTI) population. Subjects who did not have resolution of fever were censored at the time of their last non-missing post-baseline temperature assessment; this included 1 subject in the 'At Risk (<65 years)' group. Twelve subjects were excluded from summaries due to missing data or events resolving prior to initiation of study drug.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | At Risk (<65 Years) | Elderly (65-75 Years) | Very Elderly (>75 Years)
Number analyzed (Participants) | 22 | 14 | 4
hours | 41.5 [10.1 to 52.3] | 29.3 [15.5 to 43.8] | 9.4 [1.4 to 19.0]

4. Secondary Outcome: Time to Resolution of Influenza Symptoms
Description: Subjects were asked to provide an assessment of 7 influenza symptoms (cough, sore throat, nasal congestion, myalgia [aches and pains], headache, feverishness, and fatigue) on a 4-point severity scale (0, absent; 1, mild; 2, moderate; 3, severe) beginning at Screening then twice daily beginning on Day 1 through to Day 13, and prior to the subject's clinic visit on Day 14. Once all symptoms were scored a 0 or 1 for at least 48 hours, recordings were discontinued. The time to alleviation of symptoms, defined as the time from initiation of study drug until the start of the 21.5-hour period (24 hours less 10%), where all symptoms of influenza were recorded as none (0) or mild (1), was estimated overall and for each age group using the Kaplan-Meier method.
Time Frame: 14 days
Population: Intent to treat infected (ITTI) population. Subjects who did not experience alleviation of symptoms were censored at the date of their last non-missing post-baseline assessment; this included 5 subjects in the 'At Risk (<65 years)' group, 4 subjects in the 'Elderly (65-75 years)' group and 2 subjects in the 'Very Elderly (>75 years)' group.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | At Risk (<65 Years) | Elderly (65-75 Years) | Very Elderly (>75 Years)
Number analyzed (Participants) | 28 | 19 | 5
hours | 124.8 (10.59) | 114.5 (20.37) | 54.0 (9.45)

5. Secondary Outcome: Changes in Influenza Virus Titer in Nasopharyngeal Samples in Response to Treatment.
Description: Change in influenza viral titers was defined as the time-weighted change from Baseline in log_10 tissue culture infective dose_50 (TCID50/mL) and was summarized for each treatment group.
Time Frame: Change from baseline assessed on days 3, 7 and 14.
Population: The Intent To Treat Infected (ITTI) population included all subjects who were enrolled, received study drug, and had confirmed influenza A and/or B by PCR. Eight subjects were excluded due to a negative or missing BL titer.
Measure: Median (Full Range); unit: influenza viral titer - log10 TCID50/mL
Arm/Group | At Risk (<65 Years) | Elderly (65-75 Years) | Very Elderly (>75 Years)
Number analyzed (Participants) | 27 | 15 | 2
influenza viral titer - log10 TCID50/mL
  Baseline | 4.50 [1.00 to 6.50] | 4.45 [1.25 to 6.45] | 4.70 [3.45 to 5.95]
  Day 3 - Change from baseline: number analyzed (Participants) | 26 | 7 | 0
  Day 3 - Change from baseline | -3.25 [-5.00 to 3.50] | -3.00 [-5.25 to 1.25] |
  Day 7 - Change from baseline: number analyzed (Participants) | 25 | 4 | 0
  Day 7 - Change from baseline | -4.00 [-6.00 to -0.50] | -2.13 [-3.75 to -0.75] |
  Day 14 - Change from baseline: number analyzed (Participants) | 24 | 3 | 0
  Day 14 - Change from baseline | -3.88 [-6.00 to -0.50] | -3.25 [-3.75 to -0.75] |

6. Secondary Outcome: Time to Reduction in Viral Shedding
Description: Assessment of viral shedding in bilateral, mid-nasal swab specimens taken at baseline and then on Day 3, 7 and 14.
Time Frame: 14 days
Population: Intent to treat infected (ITTI) population + ITT population with positive baseline influenza viral titers [> 0.5 log10 TCID50/mL]. Eight subjects were excluded due to a negative or missing Baseline titer.
Measure: Count of Participants; unit: Participants
Arm/Group | At Risk (<65 Years) | Elderly (65-75 Years) | Very Elderly (>75 Years)
Number analyzed (Participants) | 27 | 15 | 2
Participants
  Baseline | 27 | 15 | 2
  Day 3: number analyzed (Participants) | 26 | 7 | 0
  Day 3 | 13 | 4 | 0
  Day 7: number analyzed (Participants) | 25 | 4 | 0
  Day 7 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 24 | 3 | 0
  Day 14 | 0 | 0 | 0

7. Secondary Outcome: Incidence of Influenza-related Complications
Description: Study personnel evaluated the subject at Screening and Days 3, 7, and 14 for the presence of clinical signs and/or symptoms of the following influenza-related complications: Sinusitis, Otitis media, Bronchitis & Pneumonia. Note that subjects with clinical signs and/or symptoms consistent with bacterial infections, including otitis media, bronchitis, sinusitis, and/or pneumonia at Screening, were not eligible for enrollment in this study. If an influenza-related complication was suspected, then a targeted physical examination was to be conducted to confirm the presence or absence of the influenza-related complication.
Time Frame: 14 days
Population: Intent-to-treat infected (ITTI) population
Measure: Number; unit: participants
Arm/Group | At Risk (<65 Years) | Elderly (65-75 Years) | Very Elderly (>75 Years)
Number analyzed (Participants) | 28 | 19 | 5
participants
  Otitis | 1 | 0 | 0
  Sinusitis | 0 | 1 | 0
  Bronchitis | 2 | 2 | 0
  Pneumonia | 0 | 1 | 0

8. Secondary Outcome: Time to Return to Usual Activities
Description: The ability to perform usual daily activities was assessed on a VAS (Visual Analogue Scale), where 0 indicates "unable to perform usual activities at all" and 10 indicates "able to perform usual activities.". The time to return to usual activities was the number of days from initiation of study drug until the subject recorded a rating of 10 (able to perform all usual activities fully) on the VAS; this was estimated for each age group and overall using the Kaplan-Meier method.
Time Frame: 14 days
Population: Subjects who did not return to normal activities were censored at the time of their last non-missing post-baseline assessment; this included 9 subjects in the 'At Risk (<65 years)' group, 12 subjects in the 'Elderly (65-75 years)' group and 2 subjects in the 'Very Elderly (>75 years)' group. Two subjects were excluded from summaries due to missing data or events resolving prior to initiation of study treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | At Risk (<65 Years) | Elderly (65-75 Years) | Very Elderly (>75 Years)
Number analyzed (Participants) | 27 | 19 | 4
days | 10.0 (0.59) | 12.1 (0.91) | 9.8 (2.76)

ADVERSE EVENTS:
Time Frame: Reports of AEs were to be collected from the time the subject signed the informed consent through to the follow-up period ending on Day 14.
Description: Adverse events were graded through use of the Division of Acquired Immune Deficiency Syndrome (DAIDS) Tables for Grading Adult and Pediatric Adverse Experiences. Influenza-related complications were not considered AEs unless they met the criteria for an SAE.
Arm/Group | At Risk (<65 Years) | Elderly (65-75 Years) | Very Elderly (>75 Years)
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/25 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/25 | 0/7
Other Adverse Events (participants affected / at risk) | 17/41 | 9/25 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | At Risk (<65 Years) (N=41) | Elderly (65-75 Years) (N=25) | Very Elderly (>75 Years) (N=7)
Breath sounds abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Carbon dioxide decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Nitrite urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT02635724/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT02635724/SAP_001.pdf